CLINICAL TRIAL: NCT07393906
Title: Eat Right, Screen Right: A Web-based, Self-paced Nutrition Risk Module and Cancer Prevention Resource
Brief Title: Colorectal Cancer Prevention Research Study: Eat Right, Screen Right
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202501397
Record Dates: First submitted 2026-01-14; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer Prevention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Eat Right, Screen Right Extension program aims to help adult learners manage nutrition risks and screening options for colorectal cancer prevention. Participants navigate through 6 tailored lessons covering user-identified, evidence-based information relevant to reducing colorectal cancer risk. First, participants receive an overview of colorectal cancer screening guidelines (e.g., age, modalities), personalized nutrition risk factors (e.g., how their intake of red meat, processed meat, and alcohol aligns with nutrition guidelines for colorectal cancer prevention), and additional optional colorectal cancer prevention topics via a branched conversational pathway selected by the participant. Subsequently, participants also have the opportunity to access five additional modules, providing more in-depth information. Self-reported outcomes include changes in cancer information overload, dietary intentions, and cancer screening intentions. This is an extension of previously funded pilot study and aims to enhance reach by leveraging the UF/IFAS Extension infrastructure allowing participants to achieve the following goals: (1) demonstrate accurate understanding of the modifiable dietary behavior that decrease colorectal cancer risk, (2) demonstrate understanding of screening guidelines and several ways to screen for colorectal cancer (e.g., home stool tests, colonoscopy, others), (3) develop confidence to obtain colorectal cancer screening and stay up to date with screening based on guidelines, (4) apply behavior change strategies to support cancer prevention behaviors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to understand English
* Access to a computer or mobile device

Exclusion Criteria:

* 17 years or younger
* Unable to understand English
* No access to a computer or mobile device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All populations welcome.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Intentions to obtain colorectal cancer screening | From enrollment up to 24 months. If, within 8 weeks of enrollment, participants have not completed the self-paced intervention, a reminder to complete the intervention/post-evaluation will be sent via email.
  Two self-report questionnaire measures on a 7-point Likert scale, where 1 = strongly disagree and 7 = strongly agree (i.e., I want to get screened for colorectal cancer, I plan to talk to my doctor about colorectal cancer)." On the 7-point Likert scale, higher scores would indicate stronger intentions to screen. We also ask one question about screening intentions/readiness with response options: a) I am not planning to screen in the next 6 months, b) I am thinking about screening, but not in the next 6 months, c) I am considering screening in the next 6 months, d) I am already taking steps to screen in the next 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University Florida - Online Study, Gainesville, Florida, United States